CLINICAL TRIAL: NCT01750021
Title: Comparison of Two Weight Reducing Diets in Obese Men
Brief Title: Effects of Fat and Carbohydrates in Obese Men
Acronym: FATFUNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011/2282
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Steatosis
MeSH Terms: conditions — Obesity; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat low carbohydrate diet (Experimental): High fat low carbohydrate diet
  Interventions: Dietary Supplement: High fat low carbohydrate diet
- Low fat high carbohydrate diet (Experimental): Low fat high carbohydrate diet
  Interventions: Dietary Supplement: Low fat high carbohydrate diet

INTERVENTIONS:
Dietary Supplement: High fat low carbohydrate diet — 70E% fat, 20E% protein, 10E% carbohydrates
  Arms: High fat low carbohydrate diet
Dietary Supplement: Low fat high carbohydrate diet — 20E% fat, 20E% protein, 60E% carbohydrates
  Arms: Low fat high carbohydrate diet

SUMMARY:
Obesity has become a global epidemic, and treating and preventing obesity appears to be one of the world's greatest challenges. The disorder is associated with a wide range of metabolic and hormonal changes, including the development of insulin resistance, changes in adipose tissue function, increased levels of blood lipids, cardiovascular disease and obesity induced fatty liver. Obesity is characterized by inflammation in adipose tissue, altered fat storage capacity and increased exchange of lipids between adipose tissue and blood, and increased secretion of cytokines from adipose tissue. Cytokines are believed to play a central role in the regulation of adipose tissue, the size of adipocytes and other metabolic conditions.

The hepatic synthesis of lipoproteins and interaction with adipose tissue is essential for the body's energy storages. The central role of the liver in energy supply, fat storage and normalization of blood values implies the importance of investigating the interaction between adipose tissue and liver to increase knowledge about the morbidity of obesity. Central obesity and insulin resistance are clear risk factors for the development of fatty liver, but the importance of diet is unclear. The common perception is that fatty liver condition can be improved by a reduction in dietary fat and cholesterols, but the relationship is unclear, and contradictory findings occur in epidemiological studies. It is therefore necessary to better understand the impact of the different macro-nutrients.

The purpose of this study is to determine whether two weight reducing diets with equal calorie levels that contain high or low fat differentially affects the adipose tissue function, distribution of body fat, as well as tissue, blood and urine levels of inflammatory markers, lipids, vitamins, hormones and other substances that may be related to metabolically health.

ELIGIBILITY:
Inclusion Criteria.

* Healthy men.
* BMI 30-40.
* Fasting blood glucose < 7 mM.
* Stable body weight last 2 months.

Exclusion Criteria.

* High intake of alcohol.
* Medication affecting glucose or lipid metabolism.
* Allergy towards important food items in the diet.
* Inflammatory bowel disease.
* Surgery or use of antibiotics last 2 months.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in adipose tissue | Baseline and 3 months and 6 months
  CT, body composition, molecular analyses of adipose tissue

SECONDARY OUTCOMES:
Changes in metabolic parameters | Baseline and 3 months and 6 months
  Molecular and biochemical analyses of tissue, blood and urine
Changes in inflammatory parameters | Baseline and 3 months and 6 months
  Molecular and biochemical analyses of tissue, blood and urine
Changes in endocrine parameters | Baseline and 3 months and 6 months
  Molecular and biochemical analyses of tissue, blood and urine
Changes in metabolic health | Baseline and 3 months and 6 months
  Clinical and biochemical data
Changes in adipose tissue distribution | Baseline and 3 months and 6 months
  Evaluation of adipose tissue distribution by CT
Changes in steatosis | Baseline and 3 months and 6 months
  Evaluation by CT

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Mellgren, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Veum VL, Laupsa-Borge J, Eng O, Rostrup E, Larsen TH, Nordrehaug JE, Nygard OK, Sagen JV, Gudbrandsen OA, Dankel SN, Mellgren G. Visceral adiposity and metabolic syndrome after very high-fat and low-fat isocaloric diets: a randomized controlled trial. Am J Clin Nutr. 2017 Jan;105(1):85-99. doi: 10.3945/ajcn.115.123463. Epub 2016 Nov 30. PMID 27903520